CLINICAL TRIAL: NCT06190236
Title: Integration of Neurofunctional Phenotyping Into a Preliminary Investigation of Stand-alone Web-based Cognitive Behavioral Therapy (CBT4CBT) for Alcohol Use Disorder
Brief Title: Integration of Neurofunctional Phenotyping Into Investigation of CBT4CBT for AUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20026419
Record Dates: First submitted 2023-11-20; First posted 2024-01-05 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Alcohol Abuse; Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — WW Domain-Containing Oxidoreductase; Ethanol

STUDY DESIGN:
Intervention Model Description: There will be two arms, one a control and the other arm utilizing a stand-alone web-based cognitive behavioral therapy (CBT4CBT) for alcohol use disorder. This study will utilize a 3:1 randomization favoring intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): This arm with utilize a stand-alone web-based cognitive behavioral therapy (CBT4CBT) for alcohol use disorder
  Interventions: Behavioral: Stand-alone web-based cognitive behavioral therapy (CBT4CBT) for alcohol use disorder
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Stand-alone web-based cognitive behavioral therapy (CBT4CBT) for alcohol use disorder — CBT4CBT is a 7-module web-delivered program based on CBT, an evidence-based behavioral treatment for alcohol use disorder (AUD).
  Arms: Experimental

SUMMARY:
Alcohol use and misuse are prevalent in the United States. Alcohol use disorder (AUD) is the most common substance use disorder. Evidence-based treatments are effective; however, most people with AUD do not receive treatment, and among those who do, responses to treatment modalities vary. Technology provides the opportunity to expand treatment and improve outcomes. Therefore, the overall goal of this project is to incorporate neurofunctional phenotyping into a preliminary investigation of the feasibility of providing mobile CBT4CBT for AUD among a non-treatment seeking population

DETAILED DESCRIPTION:
Nationally, alcohol is the third leading preventable cause of death. In 2019, 14.1 million adults had an alcohol use disorder (AUD). However, most people with AUD do not receive treatment, and treatments are only moderately effective among those who do receive treatment largely due to the heterogeneity of people with AUD. Precision medicine is a method to guide tailoring individual treatment regimens and improve outcomes in evidence-based treatments. Recently, neurofunctional phenotyping approaches have emerged as a promising avenue to advance precision medicine in AUD. For example, studies of the Addictions Neuroclinical Assessment (ANA) framework-a neuroscience-based framework that uses three neurofunctional domains that are considered critical to the development and maintenance of AUD-suggest there are associations between ANA domains and drinking behavior. However, the utility of phenotyping approaches has not been investigated in behavioral treatment modalities for AUD. Additionally, although AUD is the most common substance use disorder (SUD), fewer people in need of AUD treatment receive it compared to treatment for other use disorders. Many of these individuals, particularly those with mild AUD, can reduce or cease alcohol use without specialized treatment. However, efforts to refer those with more severe AUD to community residential or outpatient programs have been largely unsuccessful, especially among women who often face practical barriers like lack of transportation and childcare. Technology offers innovative opportunities to make treatment more readily accessible to those in need. Computer-Based Training for Cognitive Behavioral Therapy (CBT4CBT) is a web-based intervention with demonstrated effectiveness as an adjunct to standard AUD and other drug use disorder treatment programming. To-date, however, it has not been tested with non-treatment seeking men and women with AUD. For the proposed study, a sample of non-treatment seeking people with AUD will be recruited using ResearchMatch.org and randomized (3:1) to complete the mobile CBT4CBT program or an assessment only control condition stratified by sex (N=248 total; females: n=93 CBT4CBT, n=31 Control; males: n=93 CBT4CBT, n=31 Control). Feasibility and acceptability of CBT4CBT will be assessed among participants in the CBT4CBT condition. Study assessments that include self-reported AUD outcomes and neurofunctional assessments will be administered to all participants at baseline, immediately post-intervention, and at one month following the intervention period. All outcomes will also be assessed for sex differences using sex-stratified analyses.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* Male or female sex assigned at birth
* Meet DSM-5 Alcohol Use Disorder criteria
* report recent heavy alcohol use during the past month
* access to a smart mobile device or computer
* English-speaking.
* We are not excluding any participants based on gender identity.

Exclusion Criteria:

* currently receiving specialized professional SUD treatment
* presenting with language barriers, cognitive impairment, or serious medical or psychiatric illness that would preclude them from providing informed consent or participating in the ResearchMatch.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
Examine feasibility of CBT4CBT use as a mobile stand-alone intervention in a sample of non-treatment seeking people with AUD | 4 week check in and follow-up visit 1 (immediately after 8 week intervention period ends)
  Use of mobile CBT4CBT outside of specialized SUD treatment settings will be feasible for participants, as measured by participants completing a mean number of 70% of modules within the 8-week CBT4CBT intervention period. The outcome variable will be the mean number of modules completed (out of 7).
Examine the acceptability of CBT4CBT as a mobile stand-alone intervention in a sample of non-treatment seeking people with AUD | 4 week check in and follow-up visit 1 (immediately after 8 week intervention period ends)
  Use of mobile CBT4CBT outside of specialized SUD treatment settings will be acceptable for participants measured by 80% of participants reporting they are satisfied with CBT4CBT program. The outcome variable will be the mean satisfaction rating based on the following question: Overall, how satisfied are you with the intervention you received? (1, very dissatisfied to 5, very satisfied).

SECONDARY OUTCOMES:
Assess AUD outcomes (absence of heavy drinking days) utilizing the Timeline Follow Back (TLFB) in a sample of non-treatment seeking people with AUD who have access to the CBT4CBT compared to those who do not | Follow-up study visit 1 (immediately after intervention period and follow-up study visit 2 (one month later)
  Participants in the CBT4CBT condition will be less likely to report any heavy drinking days during the last month of the intervention period and during the month following the end of the intervention than those in the control condition based on the TLFB. The TLFB measures the quantity and frequency of past month alcohol use. The outcome variable will be absence of heavy drinking days (yes/no).
Assess AUD outcomes (recovery total score) utilizing the Substance USe Recovery Evaluator (SURE) in a sample of non-treatment seeking people with AUD who have access to the CBT4CBT compared to those who do not | Follow-up study visit 1 (immediately after intervention period and follow-up study visit 2 (one month later)
  Participants in the CBT4CBT condition will report higher total scores on the SURE during the last month of the intervention period and during the month following the end of the intervention than those in the control condition based on the TLFB. The SURE is a 21-item measure of holistic recovery. Total scores range from 21 to 63 with higher scores indicating better recovery. The outcome variable will be the total score on the SURE.
Evaluate sex differences in feasibility of CBT4CBT use as a mobile stand-alone intervention in a sample of non-treatment seeking people with AUD | 4 week check in and follow-up visit 1 (immediately after 8 week intervention period ends)
  In the CBT4CBT condition, females will complete more CBT4CBT on average than males. The outcome variable will be the mean number of modules completed (out of 7).
Evaluate sex differences in the acceptability of CBT4CBT as a mobile stand-alone intervention in a sample of non-treatment seeking people with AUD | Baseline, Follow-up study visit 1 (immediately after intervention period) and follow-up study visit 2 (one month later)
  In the CBT4CBT condition, females will report higher mean satisfaction ratings for CBT4CBT than males. The outcome variable will be the mean satisfaction rating based on the following question: Overall, how satisfied are you with the intervention you received? (1, very dissatisfied to 5, very satisfied).
Evaluate sex differences in AUD outcomes (absence of heavy drinking days) utilizing the Timeline Follow Back (TLFB) in a sample of non-treatment seeking people with AUD who have access to the CBT4CBT compared to those who do not. | Last month of the intervention and one month following the end of the intervention
  Participants in the CBT4CBT condition will be less likely to have any heavy drinking days than the control group during the last month of the intervention period and during the month following the end of the intervention for both males and females.
Evaluate sex differences in AUD outcomes (recovery total score) utilizing the Substance USe Recovery Evaluator (SURE) in a sample of non-treatment seeking people with AUD who have access to the CBT4CBT compared to those who do not. | Last month of the intervention and one month following the end of the intervention
  Participants in the CBT4CBT condition will have higher recovery scores based on the SURE than the control group during the last month of the intervention period and during the month following the end of the intervention for both males and females.
Examine associations between ANA neurofunctional and social domains at baseline | Last month of the intervention and one month following the end of the intervention
  Associations between domains and absence of heavy drinking days (yes/no) during the last month of the intervention period and during the month following the end of the intervention will vary by domain (i.e., negative emotionality, incentive salience, executive function, and social environment). Domains will be assessed using the ANA Domains Brief Scale (ANA Brief, 15-items, higher scores indicate greater impairment) and the Health Leads Social Needs Survey (HLSN, 8-items, higher scores indicate greater impairment).
Examine absence of heavy drinking days after access to the CBT4CBT program in a sample of non-treatment seeking people with AUD. | Last month of the intervention and one month following the end of the intervention
  Associations between domains and absence of heavy drinking days (yes/no) during the last month of the intervention period and during the month following the end of the intervention will vary by domain (i.e., negative emotionality, incentive salience, executive function, and social environment)

CONTACTS AND LOCATIONS:
Overall Officials: Dace Svikis, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No